CLINICAL TRIAL: NCT04221542
Title: A Phase 1 Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of AMG 509 in Subjects With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Study of AMG 509 in Participants With Metastatic Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: BeiGene (Industry); BeOne (China only) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20180146; 2023-504361-23 (Other: EU CT Number)
Record Dates: First submitted 2019-12-16; First posted 2020-01-09 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: AMG 509; mCRPC; Metastatic Castration-resistant Prostate Cancer; Prostate cancer; PSMA; STEAP1; STEAP1 targeted therapy; Solid tumor; Immunotherapy; Immuno-oncology; Immunooncology; Bispecific T-Cell engager®; BiTE®; XmAb®
MeSH Terms: conditions — Prostatic Neoplasms; Bites and Stings | interventions — abiraterone; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1: AMG 509 Intravenous (IV) Monotherapy (Experimental): Part 1 will evaluate AMG 509 in participants with metastatic castration-resistant prostate cancer (mCRPC) who have been previously treated with novel hormonal therapy (NHT) and 1 to 2 prior taxanes.
  The dose exploration phase of the study will estimate the maximum tolerated dose (MTD) of AMG 509 using a Bayesian logistic regression model (BLRM; Neuenschwander et al, 2008).
  Recommended phase 2 dose (RP2D) may be identified based on emerging safety, efficacy, PK, and pharmacodynamics (PD) data, as well as patient experience prior to reaching an MTD. Alternative dosing schedule(s) (including a third step dose) may be explored based on emerging efficacy, safety, PK data and patient experience.
  During the dose-expansion phase, individual cohorts of participants from China will be enrolled with a safety lead-in at 1 dose level below the MTD or RP2D followed by evaluation at the MTD or RP2D to confirm the safety, tolerability, MTD and/or RP2D of AMG 509 in Chinese participants.
  Interventions: Drug: AMG 509
- Part 2: AMG 509 Subcutaneous (SC) Monotherapy (Experimental): Part 2 will explore the safety, tolerability, and PK of AMG 509 SC dosing in participants with mCRPC who have been previously treated with NHT and 1 to 2 prior taxanes.
  Recommended phase 2 dose for SC monotherapy may be identified based on emerging safety, efficacy, PK, and PD data, as well as patient experience prior to reaching an MTD.
  Interventions: Drug: AMG 509
- Part 3: AMG 509 IV Monotherapy in Earlier Lines of Treatment (Experimental): Part 3 will explore AMG 509 in participants with mCRPC who have received no, or 1-2 prior NHTs (may have been given for hormone-sensitive prostate cancer [HSPC]) and no prior taxanes (unless administered in HSPC setting). This dose-expansion will be conducted to confirm safety, PK, and PD of AMG 509 at the MTD or RP2D determined in Part 1 dose exploration, and to obtain further safety and efficacy data and correlative biomarker analysis.
  Interventions: Drug: AMG 509
- Part 4: AMG 509 IV Combination Therapy (Experimental): Part 4 will explore the safety, tolerability, and PK of AMG 509 for participants with mCRPC who have received no or 1 to 2 prior NHTs given in any disease setting depending on the part (dose-expansion phase: prior therapies including at least 1 prior NHT and either 0 or 1 prior poly-ADP ribose polymerase [PARP] inhibitor), at dose regimens previously determined to be safe and tolerable in Part 1, in combination with abiraterone acetate (Part 4A) or enzalutamide (Part 4B) and no or 1 prior taxane for hormone sensitive disease in Parts 4A and 4B.
  Interventions: Drug: AMG 509; Drug: Abiraterone; Drug: Enzalutamide
- Part 5: AMG 509 IV Monotherapy in Outpatient Setting (Experimental): Part 5 will evaluate the safety and tolerability of AMG 509 IV dosing in participants with mCRPC who have been previously treated with NHT and 1 to 2 prior taxanes, when administered in outpatient infusion centers.
  The Part 5 dosing regimen and schedule was selected based on emerging data and dose level review team (DLRT) recommendations and will utilize the doses explored in Part 1 dose-expansion phase.
  Interventions: Drug: AMG 509
- Part 6: AMG 509 IV as Monotherapy and Combination Therapy With Abiraterone Acetate (Experimental): Part 6 will evaluate the preliminary efficacy, safety, tolerability, and PK of AMG 509 (alone or in combination with abiraterone acetate) for participants with mCRPC who have progressed on only 1 prior NHT (prior exposure to ≤ 6 cycles of taxane is allowed in mHSPC setting) and who have Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 measurable disease.
  Part 6 dosing regimen has been previously determined as safe and tolerable and is aligned with the dosing schedule for Parts 3 and 4A expansion.
  Interventions: Drug: AMG 509; Drug: Abiraterone
- Part 7 (China only): AMG 509 IV as Monotherapy or in Combination With Abiraterone Acetate (Experimental): Part 7 will only include participants from China. This part will evaluate safety and tolerability of AMG 509 IV dosing in participants who have been previously treated with NHT and 1 to 2 prior taxanes.
  Part 7 dosing regime will first be enrolled to dose level-1 (1.0 mg target dose) and if tolerated and if DLRT determines it is safe to escalate to the MTD/RP2D, 1.5 mg every 2 weeks (Q2W) dosing regimen may be explored. If the RP2D is safe and tolerable and once AMG 509 monotherapy dose confirmation is complete, a cohort of participants to receive AMG 509 combination therapy with abiraterone acetate may be initiated.
  Interventions: Drug: AMG 509; Drug: Abiraterone

INTERVENTIONS:
Drug: AMG 509 — AMG 509 administered as an IV infusion (Parts 1, 3, 4 and 5) or SC injection (Part 2).
  Other Names: xaluritamig
Drug: Abiraterone — Abiraterone administered as oral tablets.
  Arms: Part 4: AMG 509 IV Combination Therapy; Part 6: AMG 509 IV as Monotherapy and Combination Therapy With Abiraterone Acetate; Part 7 (China only): AMG 509 IV as Monotherapy or in Combination With Abiraterone Acetate
Drug: Enzalutamide — Enzalutamide administered as oral tablets.
  Arms: Part 4: AMG 509 IV Combination Therapy

SUMMARY:
The overall aim of the trial is to evaluate the safety, tolerability, and pharmacokinetics (PK) of AMG 509 (monotherapy and in combination with abiraterone acetate and enzalutamide) and to evaluate preliminary efficacy. As of Protocol Amendment 10 (09 July 2025), only Parts 4A expansion, 6, and 7 are open to accrual.

ELIGIBILITY:
Inclusion Criteria:

* Parts 1, 2, 5 and 7: Participants with histologically or cytologically confirmed metastatic castration-resistant prostate cancer (mCRPC) who are refractory to a novel antiandrogen therapy (abiraterone acetate and/or enzalutamide, apalutamide, or darolutamide) and have failed at least 1 (but not more than 2) taxane regimens including for metastatic hormone-sensitive prostate cancer (mHSPC) (or who are deemed medically unsuitable to be treated with a taxane regimen or have actively refused treatment with a taxane regimen). Note: A taxane regimen is defined as a minimum exposure of 2 cycles of a taxane. Any NHT that has been administered and has been stopped for reasons other than progression will not be counted as an additional line of treatment.

  1. Dose exploration phase: Novel antiandrogen therapy must have been given for treatment of metastatic disease.
  2. Dose-expansion phase: participants must not have had more than 2 NHTs and 2 taxane regimens in any setting, and an additional up to 2 other systemic anti-cancer treatments are allowed (eg, anti-PD1, PARP inhibitors, radioligand therapies, sipuleucel-T, experimental agents) Note: Combinations are considered one systemic anti-cancer treatment.
* Part 3: Participants with histologically or cytologically confirmed mCRPC who have received no or 1-2 prior NHTs (abiraterone acetate, enzalutamide, apalutamide, or darolutamide) given in any disease setting and who are deemed medically unsuitable to be treated with a taxane regimen or have actively refused treatment with a taxane regimen (unless taxane treatment was administered in HSPC setting). 0 1 prior PARP inhibitors or sipuleucel-T treatments are acceptable. Participants who received prior investigational therapy for the treatment of metastatic disease are not eligible.
* Parts 4A, 4B and 7:

  1. Participants with histologically or cytologically confirmed mCRPC who have received no or 1-2 prior NHTs (given in any disease setting depending on the part), and no or 1 taxane regimen (for HSPC).
  2. Dose-expansion phase: at least 1 prior NHT must have been given; 0-1 prior PARP inhibitors are acceptable.
  3. 4A: Participants planning to receive abiraterone acetate for the first time (participants who received prior abiraterone acetate are not eligible). Participants may have had exposure to up to 2 NHTs with a similar mechanism of action (apalutamide, enzalutamide or darolutamide) in the non-mCRPC and mCRPC setting.
* Dose-expansion phase: up to approximately 10 participants with prior exposure to abiraterone acetate may be enrolled into Part 4A expansion cohort.

  d. 4B: Participants planning to receive enzalutamide for the first time (participants who received prior enzalutamide/apalutamide or daralutamide are not eligible).
* Part 6:

  1. Prior disease progression on 1, and only 1, NHT (either enzalutamide, apalutamide, or darolutamide) is required. NOTE: Prior progression on or intolerance to abiraterone is not allowed.
  2. No prior treatment with any chemotherapy regimen in the mCRPC setting; ≤ 6 cycles of docetaxel treatment in the mHSPC setting is allowed.
  3. mCRPC with ≥ 1 RECIST v1.1 measurable lesion that is present on baseline computed tomography (CT) or magnetic resonance imaging (MRI).
* All parts:
* Participants must have undergone bilateral orchiectomy or be on continuous androgen-deprivation therapy with a gonadotropin releasing hormone (GnRH) agonist or antagonist.
* Total serum testosterone ≤ 50 ng/dL or 1.7 nmol/L.
* Evidence of progressive disease, defined as 1 or more Prostate Cancer Working Group 3 (PCWG3) criteria:

  1. PSA level ≥ 1 ng/mL that has increased on at least 2 successive occasions at least 1 week apart.
  2. Nodal or visceral progression as defined by RECIST v1.1 with PCGW3 modifications.
  3. Appearance of 2 or more new lesions in bone scan.
* Eastern Cooperative Oncology Group performance status of 0-1.
* Life expectancy ≥ 3 months.
* Adequate organ function, defined as follows:

  1. Hematological function:

     1. absolute neutrophil count ≥ 1 x 10^9/L (without growth factor support within 7 days from screening assessment).
     2. platelet count ≥ 75 x 10^9/L (without platelet transfusion within 7 days from screening assessment).
     3. hemoglobin ≥ 9 g/dL (90 g/L) (without blood transfusion within 7 days from screening assessment).
  2. Renal function:

     1. estimated glomerular filtration rate based on Modification of Diet in Renal Disease calculation ≥ 30 ml/min/1.73 m^2.
  3. Hepatic function:

     1. aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x upper limit of normal (ULN) (or < 5 x ULN for participants with liver involvement).
     2. total bilirubin (TBL) < 1.5 x ULN (or < 2 x ULN for participants with liver metastases).
  4. Cardiac function:

     1. left ventricular ejection fraction > 50% (2-D transthoracic echocardiogram [ECHO] is the preferred method of evaluation; multi-gated acquisition scan is acceptable if ECHO is not available).
     2. Baseline electrocardiogram (ECG) QTcF ≤ 470 msec (average of triplicate values).
  5. Pulmonary function:

     1. baseline oxygen saturation > 92% on room air at rest and no oxygen supplementation.

Part 3-Retreatment group:

* Deriving benefit from initial treatment with AMG 509 as evidenced by one of the following:

  1. confirmed PSA50 response.
  2. radiographic stable disease/partial response/complete response during 6 cycles of initial treatment with AMG 509 and without progression during the first 6 cycles.
* No discontinuation for toxicity during the initial treatment with 6 cycles of AMG 509.
* Progressive disease as defined in I106 within 12 months of final dose in their initial treatment with 6 cycles (EOT_1).
* Willingness to have a fresh tumor biopsy prior to initiating the additional course of treatment, depending on safety and feasibility as assessed by investigator.

Key Exclusion Criteria:

* Pathological finding consistent with pure small cell, neuroendocrine carcinoma of the prostate or any other histology different from adenocarcinoma.
* Radiation therapy within 4 weeks of first dose (or local or focal radiotherapy within 2 weeks of first dose).
* Untreated central nervous system (CNS) metastases or leptomeningeal disease. Participants with a history of treated CNS metastases are eligible if there is radiographic evidence of improvement upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study.
* Prior major surgery within 4 weeks of first dose.
* Participants with symptoms and/or clinical signs and/or radiographic signs that indicate an acute and/or uncontrolled active systemic infection within 7 days prior to the first dose of investigational product administration. Simple urinary tract infections and uncomplicated bacterial pharyngitis are permitted if responding to active treatment and after consultation with sponsor. Screening for chronic infectious conditions is not required.
* Confirmed history or current autoimmune disease or other diseases resulting in permanent immunosuppression or requiring permanent immunosuppressive therapy.
* History of arterial or venous thrombosis (eg, stroke, transient ischemic attack, pulmonary embolism, or deep vein thrombosis); for arterial thrombosis within 12 months of AMG 509 initiation; for venous thrombosis, 6 months and stable on anti-coagulation. Participants with a recent history of venous thrombosis must be maintained on the same anti-coagulation therapy for a minimum of 28 days prior to first dose of study treatment.
* Myocardial infarction and/or symptomatic congestive heart failure (New York Heart Association > class II) within 12 months of first dose of AMG 509 with the exception of ischemia or non-ST segment elevation myocardial infarction controlled with stent placement and confirmed by a cardiologist more than 6 months prior to first dose of AMG 509.
* Any anti-cancer therapy or immunotherapy within 4 weeks of start of first dose, not including luteinizing hormone-releasing hormone (LHRH)/GnRH analogue (agonist/antagonist).
* Prior prostate specific membrane antigen (PSMA) radionuclide therapy within 2 months prior to AMG 509 unless participant received < 2 cycles (Note: a participant cannot have received PSMA radionuclide therapy < 35 days prior to enrollment if 1 cycle was given). Parts 3 and 4: prior PSMA radionuclide therapy is prohibited. Participants on a stable bisphosphonate or denosumab regimen for ≥ 30 days prior to enrollment are eligible (exception: part 3 retreatment).
* Part 3-Retreatment only: Any anti-cancer therapy or immunotherapy, not including luteinizing hormone-releasing hormone/gonadotropin releasing hormone (LHRH/GnRH) analogue (agonist/antagonist), and/or bisphosphonate or denosumab regimen after last dose of AMG 509 initial course of treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 479 (Estimated)
Dates: Start 2020-03-04 (Actual); Primary Completion 2030-03-22 (Estimated); Study Completion 2032-03-21 (Estimated)

PRIMARY OUTCOMES:
Parts 1-5 and 7: Incidence of Treatment-emergent Adverse Events | 3 years
Parts 1-5 and 7: Incidence of Treatment-related Adverse Events | 3 years
Parts 1-5 and 7 Dose Exploration Cohorts Only: Dose Limiting Toxicities (DLTs) | 28 days
Parts 1-5 and 7: Number of Participants with Changes in Vital Signs | 3 years
Parts 1-5 and 7: Number of Participants with Changes in Electrocardiogram (ECG) Records | 3 years
Parts 1-5 and 7: Number of Participants with Changes in Clinical Laboratory Test Results | 3 years
Part 6: Objective Response (OR) per RECIST v1.1 | 3 years

SECONDARY OUTCOMES:
Parts 1-7: Maximum Serum Concentration (Cmax) for AMG 509 | 3 years
  To characterize the pharmacokinetics (PK) of AMG 509
Parts 1-7: Time to Maximum Serum Concentration (Tmax) for AMG 509 | 3 years
  To characterize the pharmacokinetics (PK) of AMG 509
Parts 1-7: Minimum Serum Concentration (Cmin) for AMG 509 | 3 years
  To characterize the pharmacokinetics (PK) of AMG 509
Parts 1-7: Area Under the Concentration-time Curve (AUC) Over the Dosing Interval for AMG 509 | 3 years
  To characterize the pharmacokinetics (PK) of AMG 509
Parts 1-7: Accumulation Following Multiple Dosing for AMG 509 | 3 years
  To characterize the pharmacokinetics (PK) of AMG 509
Parts 1-5 and 7: OR per RECIST v1.1 | 3 years
  To evaluate preliminary anti-tumor activity of AMG 509
Parts 1-7: Prostate Specific Antigen (PSA) Response | 3 years
  To evaluate preliminary anti-tumor activity of AMG 509
Parts 1-5 and 7: PSA Decline of at Least 50% From Baseline at 12 Weeks | Week 12
  To evaluate preliminary anti-tumor activity of AMG 509
Parts 1-7: Radiographic Duration of Response (DOR) | 3 years
  To evaluate preliminary anti-tumor activity of AMG 509
Parts 1-5 and 7: PSA DOR | 3 years
  To evaluate preliminary anti-tumor activity of AMG 509
Parts 1-5 and 7: Radiographic Time to Progression | 3 years
  To evaluate preliminary anti-tumor activity of AMG 509
Parts 1-5 and 7: PSA Time to Progression | 3 years
  To evaluate preliminary anti-tumor activity of AMG 509
Parts 1-5 and 7: Radiographic Progression-free Survival (PFS) | 3 years
  To evaluate preliminary anti-tumor activity of AMG 509
Parts 1-5 and 7: PSA PFS | 3 years
  To evaluate preliminary anti-tumor activity of AMG 509
Part 6: Radiographic PFS per Prostate Cancer Working Group 3 (PCWG3)-modified RECIST v1.1 | 3 years
  To evaluate preliminary anti-tumor activity of AMG 509
Parts 1-2, 5 and 7: 6 Month Radiographic PFS | 6 months
  To evaluate preliminary anti-tumor activity of AMG 509
Part 3 and 4: 1, 2, and 3-year Radiographic PFS | Year 1, 2, and 3
  To evaluate preliminary anti-tumor activity of AMG 509
Parts 1-5: 1, 2, and 3-year Overall Survival (OS) | Year 1, 2, and 3
  To evaluate preliminary anti-tumor activity of AMG 509
Parts 1-5: Circulating Tumor Cells Response (CTC0) | 3 years
  To evaluate preliminary anti-tumor activity of AMG 509
Parts 1-5: Rate of Circulating Tumor Cells (CTC) Conversion | 3 years
  To evaluate preliminary anti-tumor activity of AMG 509
Parts 1-5: Time to Symptomatic Skeletal Events | 3 years
  To evaluate preliminary anti-tumor activity of AMG 509. Measure of disease burden based on PCWG3-recommended endpoints.
Parts 1-5: Alkaline Phosphatase (Total, Bone) | 3 years
  To evaluate preliminary anti-tumor activity of AMG 509. Measure of disease burden based on PCWG3-recommended endpoints.
Parts 1-5: Lactate Dehydrogenase (LDH) | 3 years
  To evaluate preliminary anti-tumor activity of AMG 509. Measure of disease burden based on PCWG3-recommended endpoints.
Parts 1-5: Hemoglobin | 3 years
  To evaluate preliminary anti-tumor activity of AMG 509. Measure of disease burden based on PCWG3-recommended endpoints.
Parts 1-5: Urine N-telopeptide | 3 years
  To evaluate preliminary anti-tumor activity of AMG 509. Measure of disease burden based on PCWG3-recommended endpoints.
Parts 1-5: Neutrophil-to-lymphocyte Ratio | 3 years
  To evaluate preliminary anti-tumor activity of AMG 509. Measure of disease burden based on PCWG3-recommended endpoints.
Part 6: Incidence of Treatment-emergent Adverse Events | 3 years
Part 6: Incidence of Treatment-related Adverse Events | 3 years
Part 6: Number of Participants with Changes in Vital Signs | 3 years
Part 6: Number of Participants with Changes in Clinical Laboratory Test Results | 3 years
Part 6: Disease Control per RECIST v1.1 | 3 years
Parts 6 and 7: OS | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (55):
- United States (25):
  - City of Hope National Medical Center, Duarte, California
  - Providence Saint Jude Medical Center, Fullerton, California
  - University of California San Francisco, San Francisco, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - MidAmerica Cancer Care, Merriam, Kansas
  - Tulane Medical Center, New Orleans, Louisiana
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Oncology Hematology Care Incorporated, Cincinnati, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Prisma Health Upstate, Greenville, South Carolina
  - Sanford Oncology Clinic and Pharmacy, Sioux Falls, South Dakota
  - United States Oncology Regulatory Affairs Corporate Office, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - US Oncology Research Investigational Products Center, Irving, Texas
  - Intermountain Medical Center, Murray, Utah
  - Virginia Cancer Specialists PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (2):
  - Chris OBrien Lifehouse, Camperdown, New South Wales
  - Monash Medical Centre, Clayton, Victoria
- China (5):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Fudan University Shanghai Cancer Centre, Shanghai, Shanghai Municipality
  - Zhejiang Provincial Peoples Hospital, Hangzhou, Zhejiang
- Germany (4):
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Klinikum rechts der Isar der TUM, München
  - Universitaetsklinikum Muenster, Münster
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
- Portugal (3):
  - Hospital da Luz, SA, Lisbon
  - Unidade Local de Saude de Santa Maria, EPE - Hospital de Santa Maria, Lisbon
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, EPE, Porto
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (5):
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Switzerland (4):
  - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Kantonsspital Graubuenden, Chur
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Sankt Gallen, Sankt Gallen
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital of Chang Gung Medical Foundation, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Kelly WK, Danila DC, Lin CC, Lee JL, Matsubara N, Ward PJ, Armstrong AJ, Pook D, Kim M, Dorff TB, Fischer S, Lin YC, Horvath LG, Sumey C, Yang Z, Jurida G, Smith KM, Connarn JN, Penny HL, Stieglmaier J, Appleman LJ. Xaluritamig, a STEAP1 x CD3 XmAb 2+1 Immune Therapy for Metastatic Castration-Resistant Prostate Cancer: Results from Dose Exploration in a First-in-Human Study. Cancer Discov. 2024 Jan 12;14(1):76-89. doi: 10.1158/2159-8290.CD-23-0964. PMID 37861461
- [Background] Kuipers-Connarn JN, Pourzanjani A, Bose M, Modi S, Stieglmaier J, Murphy A, Mehta K, Upreti VV. Clinical Pharmacology Characterization and Dose Selection of Xaluritamig, a Next Generation XmAb(R) 2+1 T-Cell Engager, in Prostate Cancer Patients. J Clin Pharmacol. 2025 Dec;65(12):1676-1686. doi: 10.1002/jcph.70074. Epub 2025 Aug 5. PMID 40765197
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com